CLINICAL TRIAL: NCT06671158
Title: An Evaluation of the Effectiveness and Mechanisms of Change of Measurement Based Care for Depressive and Anxiety Disorders
Brief Title: Measurement-Based Care (MBC) Implementation, Effectiveness, and Mechanisms of Change
Acronym: MBC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Virginia O'Brien, Principal Investigator, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-23-1992
Record Dates: First submitted 2024-10-10; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Depressive Disorder; Anxiety Disorders
Keywords: measurement-based care; effectiveness; RCT; implementation; psychotherapy; mechanisms of change
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Measurement-based care group (Experimental): Measurement-based care group
  Interventions: Behavioral: Psychotherapy
- Treatment-as-Usual group (Active Comparator): Treatment-as-Usual group
  Interventions: Behavioral: Psychotherapy
- Waitlist control group (No Intervention): Waitlist control group

INTERVENTIONS:
Behavioral: Psychotherapy — Individual psychotherapy for weekly 12-sessions
  Arms: Measurement-based care group; Treatment-as-Usual group

SUMMARY:
Although measurement-based care (MBC) is an evidence-based practice with known benefits, it is not always systematically implemented with fidelity. Questions remain regarding MBC's unique added value compared to usual care.

Thus, the goal of this clinical trial is to investigate the implementation outcome, effectiveness, and mechanisms of change of measurement-based care in adult behavioral health. This study implemented MBC in adult ambulatory behavioral health and will test outcomes using a pragmatic randomized control trial within the RE-AIM (Reach, Efficacy, Adoption, Implementation, and Maintenance) framework.

Researchers will compare three groups: 1) the Measurement-based care group, 2) the treatment-as-usual group, and 3) the waitlist control group. Participants will participate in weekly individual psychotherapy sessions for 12 sessions in total.

DETAILED DESCRIPTION:
Measurement-based care (MBC) is an evidenced-based practice, involving routine completion of patient-reported outcome measures and collaborative discussions between clinician and client to inform clinical decision-making and facilitate improvement. Despite its known benefits, such as reduced dropout rates and improved treatment outcomes, questions remain regarding MBC's unique effectiveness compared to standard care. Furthermore, mechanisms of change on how MBC actually works in treatment have yet to be fully investigated. Thus, the current study aims to conduct a randomized control trial to evaluate the added value of MBC, by comparing an MBC+psychotherapy group, a psychotherapy-only group, and a waitlist group with no interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Primary concern and referral reason for seeking psychotherapy are either depressive- or anxiety-related symptoms and/or psychological distress, using minimum scores as follows: PHQ-9 (score > 4), GAD-7 (score > 4), and BASE-6 (score > 18), and
2. being 18 years old or older.

Exclusion Criteria:

1. Severe physical or psychiatric conditions that would hinder the treatment (e.g., clients with acute psychosis, intellectual disability, or neurocognitive disorders who do not have the capacity to undergo informed consent and participate in the study);
2. currently receiving psychotherapy through another source;
3. significant suicidal/homicidal risk that would need immediate intervention;
4. do not have ability complete Patient-Rated Outcome Measures (PROMs) either in person or remotely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Brief Adjustment Scale-6 (BASE-6) | Completed weekly through study completion, an average of 3 to 4 months
  Self-report questionnaire designed to measure general psychological adjustment and functioning of adult-aged individuals Minimum score: 6 Maximum score: 42 A higher score indicates severe difficulty in psychological adaptation and functioning/worse outcome
Patient Health Questionnaire-9 (PHQ-9) | Completed weekly through study completion, an average of 3 to 4 months
  Evaluate depression symptoms Minimum score: 0 Maximum score: 27 A higher score indicates more severe depression/worse outcome
Generalized Anxiety Disorder-7 (GAD-7) | Completed weekly through study completion, an average of 3 to 4 months
  evaluate anxiety symptoms Minimum score: 0 Maximum score: 21 A higher score indicates more severe anxiety/worse outcome

SECONDARY OUTCOMES:
World Health Organization Quality of Life-Brief (WHOQOL-BREF) | Pre-post, through study completion, an average of 3 to 4 months
  This is a self-report measure designed to assess an individual's quality of life and well-being across four domains, including physical health, psychological well-being, social relationships, and environmental conditions Minimum score: 0 Maximum score: 100 A higher score indicates a higher quality of life/better outcome
Working Alliance Inventory-Short Form Revised (WAI-SR) | Completed monthly, through study completion, an average of 3 to 4 months
  The WAI-SR is a self-report measure of the strengths of the therapeutic alliance that clients perceive.
  Minimum score: 12 Maximum score: 60 A higher score indicates a stronger working alliance between the provider and the patient / better outcome
Vanderbilt Psychotherapy Process Scale - Patient version (VPPS) | Completed every 6 weeks; through study completion, an average of 3 to 4 months
  The VPPS-P is a patient-report measure consisting of 42 items with five subscales, including therapist exploration, negative relationship, patient psychic distress, patient participation, therapist warmth and friendliness, and patient dependency.
  Minimum score: 42 Maximum score: 210 A higher score indicates better outcome

OTHER OUTCOMES:
Clinical Global Impressions - Severity of Illness (CGI-S) | Pre-post, through study completion, an average of 3 to 4 months
  Clinical impressions of the clinician's view on the client's global functioning, the overall severity of symptoms (CGI-S) Minimum score: 1 Maximum score: 7 A higher score indicates more severe impairment/worse outcome
Patient's Global Impressions of Severity (PGI-S) | Pre-post, through study completion, an average of 3 to 4 months
  As CGI-S, the PGI-S is a 1-item global impression questionnaires that allow patients to report their own views on the severity of ongoing symptoms based on a 7-point scale Minimum score: 1 Maximum score: 7 A higher score indicates more severe impairment/worse outcome
Clinical Global Impressions - Improvement (CGI-I) | Through study completion, an average of 3 to 4 months
  Clinical impressions of the client's improvement level that the client shows throughout the therapy (CGI-I) Minimum score: 1 Maximum score: 7 A lower score indicates better outcome
Patient Global Impressions - Improvement (PGI-I) | Through study completion, an average of 3 to 4 months
  PGI-S is a 1-item global impression questionnaires that allow patients to report their own views on the response and improvement to intervention based on a 7-point scale Minimum score: 1 Maximum score: 7 A lower score indicates better outcome
Patient Attitudes with and Satisfaction towards Measurement-Based Care (PAS-MBC) | Through study completion, an average of 3 to 4 months
  A 12-item tailored questionnaire was created to fully capture clients' attitudes towards and experience with measurement-based care during their treatment.
  Minimum value: 12 Maximum value: 60 Higher score indicates better outcome/more positive attitudes toward measurement-based care

CONTACTS AND LOCATIONS:
Overall Officials: Virginia O'Brien, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Mental Health, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Due to the need to protect patient confidentiality and privacy regarding identifiable health data